CLINICAL TRIAL: NCT02406807
Title: H-reflex Responses to High-Velocity Low-Amplitude Manipulation in Adults With Chronic Non-specific Low Back Pain
Brief Title: H-reflex Responses to High-Velocity Low-Amplitude Manipulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Brasileiro de Osteopatia (Other)
Responsible Party: Principal Investigator, Sandro Groisman, PT, DO, MSc, DO, Instituto Brasileiro de Osteopatia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2015-03-18; First posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Low Back Pain
Keywords: chronic low back pain; HVLA manipulation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HVLA manipulation (Experimental): Osteopathic high velocity, and low amplitude spinal lumbar manipulation
  Interventions: Other: HVLA manipulation
- Sham Spinal lumbar manipulation (Sham Comparator): Just position in the side lying and not performed the high velocity and low amplitude
  Interventions: Other: Sham Spinal lumbar manipulation

INTERVENTIONS:
Other: HVLA manipulation — participant is laying on the left side, the practitioner stands in front of the participant's abdomen. The practitioner contacts the interspinous space of the L5-S1 level with the caudal; with the cephalic hand, the practitioner rotates the participant's upper body until a sense of tension is palpated at the L5-S1 segment. The practitioner places his cephalic hand at interspinous, brings participant's leg to a flexion and places the foot at the popliteal fossa, places the forearm at the participant's deltopectoral groove and the caudal forearm at the gluteal region. Following the participant's expiration, the practitioner brings the L5-S1 level to the restrictive barrier by rotating the trunk and hips to opposite directions.
  Arms: HVLA manipulation
Other: Sham Spinal lumbar manipulation — Sham manipulation
  Arms: Sham Spinal lumbar manipulation

SUMMARY:
High-Velocity Low-Amplitude (HVLA) manipulation is a known technique of the Osteopathic Manipulative Treatment (OMT) for somatic dysfunction (SD), and heart rate variability and H-reflex response are possible variables to assess its neurophysiological effects. Somatic dysfunction is an impairment or altered function of related components of the somatic system.

Studies show a transient attenuation of α-motor neuron excitability after HVLA manipulation in asymptomatic participants. According to studies, HVLA spinal manipulation increases joint mobility by blocking afferent impulses in the muscle spindle and the small-diameter free nerve, decreasing the γ-motor neuron activity.

DETAILED DESCRIPTION:
Osteopathic Manipulative Treatment (OMT) is a health science that addresses treatment to somatic dysfunction among other conditions. High-Velocity Low-Amplitude (HVLA) manipulation is a known technique, defined as a quick and short force applied to a segment with movement restriction.

Somatic Dysfunction (SD) is the impaired or altered function of the components of the somatic system: skeletal, articular and myofascial elements with their vascular, lymphatic and neural related structures. The palpatory diagnosis of the SD is based on the presence of any of the 4 TART (Tenderness, Asymmetry, Range of motion and Tissue texture change) criteria, taking into account the information provided about pain and discomfort.

There is no evidence to support the use of the term 'somatic dysfunction' and moreover, the diagnosis is based on palpatory skills. Therefore, the investigators chose the term Restriction of Movement (RM) to describe the subjectivity of the palpatory examination.

HVLA manipulation produces neurophysiological and mechanic effects. The mechanical effects described in the literature are: meniscoids release, intervertebral disc material and segmental adhesions. The neurophysiological effects occur through the stimulation of mechanoreceptors and nociceptors located in the paravertebral tissues, including the skin, muscles, tendons, ligaments, zygapophyseal joints and intervertebral discs. This changes the influx of sensory information into the Central Nervous System (CNS), and this effect can be measured by the H-reflex (reflex analogous to the spinal stretch reflex). Thus, this is a valuable tool in the assessment of α-motor neuron excitability.

Studies show a transient attenuation of α-motor neuron excitability after HVLA manipulation in asymptomatic participants. According to studies, HVLA spinal manipulation increases joint mobility by blocking afferent impulses in the muscle spindle and the small-diameter free nerve, decreasing the γ-motor neuron activity.

Most of the studies analyzed recruited healthy participants, and have found transient attenuation of α-motor neuron activity; but one study found that the manipulation does not affect the H-reflex in healthy participants. These authors attributed the findings to the change of position between intervention and assessment. In addition, the intervention was addressed to sacroiliac joint instead of the L5-S1 segment, as performed in other previous studies.

Another study assessed the effects of manipulation without changing participants' position, but unlike the study of Suter et al., the intervention was addressed to the lumbosacral joint (L5-S1) and they concluded that changing body position does not affect the H-reflex attenuation.

Therefore, the studies show divergent results for HVLA manipulation and H-reflex response, and to better understand the research problem, the investigators conducted a previous study in 20 healthy participants to assess the effects of HVLA manipulation on H-reflex and they found a transient H-reflex attenuation only in six participants.

These findings could have been affected by the presence of RM at the level L5-S1 and also by the presence of dysfunction of the Autonomic Nervous System (ANS), which is processed at medullar level and runs along neural pathways, similar to somatic afferent and efferent information.

To quantify ANS activity, one could use Nerve-Express - a device to assess heart rate variability based on RR (rate-rate) intervals. This method is used because of the major role the ANS plays on the cardiovascular system. Studies have shown the effects of cervical and lumbar HVLA manipulation on heart rate variability and on balancing the ANS.

ELIGIBILITY:
Inclusion Criteria:

* participants of both gender,
* aged between 20 and 50 years,
* healthy participants and
* participants diagnosed with non-specific chronic low back pain and healthy participants.

Exclusion Criteria:

* participants referring radiating pain to the lower limbs and any other symptoms compatible with nerve root entrapment, knee or hip degenerative diseases and abdominal pain
* participants from whom it was not possible to record the H-reflex and
* participants with absolute contraindication to HVLA manipulation.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
H-reflex measured by the electroneurophysiologic | Within one day
  Electroneurophysiologic

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Groisman, Ms, Principal Investigator — IBO